CLINICAL TRIAL: NCT02836522
Title: Validation of a Health-Related Symptom Index for Persons Diagnosed With and Either Treated or Monitored for Anal High-Grade Squamous Intraepithelial Lesions (HSIL)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-282
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Anal High-Grade Squamous Intraepithelial Lesions
Keywords: Health-Related Symptom Index; ANCHOR( ANal Cancer HSIL (high grade squamous intraepithelial lesions) Outcomes Research study)
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Assessment of Health-Related Quality — Demographic Questionnaire, ANCHOR HRSI, FACT-G, MDASI, Patient ECOG PS, PGIC

SUMMARY:
The purpose of this study is to finalize development of a questionnaire that measures health-related symptoms and concerns for persons diagnosed with, and either treated or monitored for, anal pre-cancer lesions.

ELIGIBILITY:
Inclusion Criteria:

* Consented to the ANCHOR trial as per self-report and by providing a valid referral code on the information sheet provided by the referring site. Both men and women from the ANCHOR trial will be recruited to this study.
* English fluent as we are only validating this measure in English at this time
* At least one month post-treatment for anal HSIL as per self-report, or if the person is in the ANCHOR trial observation arm, then at least one month post- randomization.
* Within two weeks post initial-treatment for anal HSIL on ANCHOR study or within two weeks post-randomization to ANCHOR study as per self-report.

NOTES:

* ANCHOR participants who are randomized to the treatment arm must have completed initial treatment and are within two weeks of initial treatment completion.
* ANCHOR participants who were treated initially with topical treatment are only eligible within two weeks after the last topical treatment application.
* ANCHOR participants who were treated initially with both topical and ablation treatments are eligible within two weeks of completing both treatments.
* ANCHOR participants who are randomized to the active monitoring arm are eligible if they are within two weeks of randomization

Exclusion Criteria:

* Has a scheduled ANCHOR follow-up appointment in the next two weeks as per self report. The purpose of this exclusion criterion is to minimize the impact on a participant's responses to a post-test evaluation the potential occurrence of an interim diagnosis or treatment event, or anxiety related to an upcoming medical follow-up.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participating ANCHOR sites
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
degree of test-retest reliability in the ANCHOR HRSI | 7-10 days
  measure from the initial assessment point to the 7-10 day follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Atkinson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Northwestern University, Evanston, Illinois
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - City College of New York, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York

REFERENCES:
- [Derived] Burkhalter JE, Atkinson TM, Berry-Lawhorn J, Goldstone S, Einstein MH, Wilkin TJ, Lee J, Cella D, Palefsky JM; ANCHOR HRQOL Implementation Group. Initial Development and Content Validation of a Health-Related Symptom Index for Persons either Treated or Monitored for Anal High-Grade Squamous Intraepithelial Lesions. Value Health. 2018 Aug;21(8):984-992. doi: 10.1016/j.jval.2018.01.018. Epub 2018 Apr 11. PMID 30098677
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02836522/ICF_000.pdf